CLINICAL TRIAL: NCT05840666
Title: Effects of Mulligan Sustained Natural Apophyseal Glides Versus McKenzie Method of Mechanical Diagnosis & Therapy in Patients With Non-Specific Chronic Low Back Pain
Brief Title: Mulligan Sustained Natural Apophyseal Glides Versus McKenzie Method in Patients With Non-Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayesha Jamil (Other)
Responsible Party: Sponsor-Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahsan Javed
Record Dates: First submitted 2023-04-05; First posted 2023-05-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
Keywords: Non-specific Low Back Pain; Sustained Natural Apophyseal Glide; McKenzie Method; Mechanical Diagnosis and Therapy; Range of Motion; Pain; Functional Disability; Fear Avoidance Beliefs
MeSH Terms: conditions — Low Back Pain; Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to three study arms and each study arm will be allocated a different intervention
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of the treatment group of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physical Therapy (CPT) Group (Active Comparator): Conventional Physical Therapy will consist of Therapeutic Ultrasound, Moist Heat-pack, TENS and standard exercises. Participants will receive 15 sessions of Conventional Physical Therapy (CPT) at a frequency of 5 sessions per week.
  Interventions: Other: Conventional Physical Therapy
- Conventional Physical Therapy (CPT) plus Mulligan SNAGs Group (Experimental): Besides Conventional Physical Therapy, Mulligan Mobilizations will be provided in this group. It consist of Extension SNAGS in prone, and Lumbar flexion SNAGS in sitting. The techniques will be applied in 3 sets with 10 repetitions and 60 seconds rest between sets.
  Interventions: Other: Mulligan Sustained Natural Apophyseal Glide (SNAG)
- Conventional Physical Therapy plus McKenzie MDT Group (Experimental): Along with Conventional Physical Therapy, McKenzie MDT will be be given in this group. It consist of Prone lying, Prone lying Elbow popups, Prone elbow Extension. Standing Extension, supine Both Knee to Chest, Sitting on chair with forward flexion. The techniques will be applied in 3 sets with 8-10 repetitions and 60 seconds rest between sets.
  Interventions: Other: McKenzie Method

INTERVENTIONS:
Other: Mulligan Sustained Natural Apophyseal Glide (SNAG) — Application of the MWM technique developed by Brian R. Mulligan. The clinical researcher will perform and holds sustained passive segmental glide at the target joint maintaining the slack whereas the patient will actively move in the direction of pain or stiffness. These MWM techniques when applied to spinal segments or joint is called sustained natural apophyseal glide (SNAG).
  Other Names: Mulligan Mobilization
  Arms: Conventional Physical Therapy (CPT) plus Mulligan SNAGs Group
Other: McKenzie Method — An active therapy technique involving repeated movements or sustained positions along with an educational component prescribed to the patient for of minimizing the pain and disability and increase the spinal range of motion. The method will involve the assessment of symptomatic and mechanical responses to repeated movements and sustained positions in the direction of preference. The method will be used for assessment and treatment of patients and with derangement syndrome.
  Other Names: Mechanical Diagnosis and Therapy (MDT)
  Arms: Conventional Physical Therapy plus McKenzie MDT Group
Other: Conventional Physical Therapy — It includes usual physical therapy care such as Therapeutic Ultrasound, Moist Heat-pack, TENS and standard exercises.
  Arms: Conventional Physical Therapy (CPT) Group

SUMMARY:
Low back pain (LBP) is the most frequent complaint encountered in clinical practice. Exercises and manual therapy prescription are common physical therapy treatments prescribed for the patients presenting with chronic low back pain. The interventions will establish the future direction for practitioners in choosing the manual therapy or repeated exercises as effective prescription and provide a basis for future research

DETAILED DESCRIPTION:
A variety of treatment interventions, modalities and techniques are used in physical therapy management of non-specific low back pain including manual therapy, exercises, neural mobilizations, stretching soft tissue techniques and dry needling etc. Out of these more recent literature supports manual therapy, self exercises, patient counseling and awareness have been recommended in back pain management guidelines, in the United States and is also frequently used in clinical practice in various countries.

Despite multiple theoretical frame works proposing the role of SNAGs and MDT mobilizations and exercises respectively, the literature on the true mechanism of direct or indirect physiological effects of these on performance or performance-related outcomes is vague and lacks justifiable procedural rigor.

The results of this study will provide information regarding the direction for practitioners in choosing the manual therapy or repeated exercises as effective prescription and provide a basis for future research.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Both genders
* Adult patents between the 20 to 45 years of age with chronic non-specific low back pain.
* Pain intensity of at least 3 or greater on 0-10 Numeric Rating Scale.
* Modified Low Back Pain Disability Questionnaire score equal to or greater than 20%.

Exclusion Criteria:

* Serious underlying pathology with red flags.
* Patients having contraindication to physical exercises.
* Females with high parity.
* Pregnant or lactating females.
* Patients who participated in any type of rehabilitative training or exercise program for back pain in last 1 month.
* Spinal deformity or Spinal stenosis.
* History of fall or trauma to spine in last one year.
* History of spinal, abdominal or hip surgery.
* Signs of nerve root compression with sensory, motor or deep tendon reflexes deficit.
* Serious underlying pathology with red flags.
* Systemic disease e.g., cardiovascular, metabolic or central nervous system.
* Osteopenia, osteoporosis.
* Medication's history (steroids, immunosuppressants, chemotherapy)
* Limb length discrepancy.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be recorded as baseline at the time of recruitment and change in pain intensity will be observed at follow up at the end of 3rd week of treatment.
  Level of pain intensity will be measured using Numeric Rating Scale. The 11-point numeric scale ranges from '0' representing no pain to '10' representing the extreme pain
Lumbar Range of Motion | Lumbar Range of Motion will be observed as baseline at the time of recruitment and change in ROM will be observed at follow up at end of 3rd week of treatment.
  Lumbar Range of motion will be measured using inclinometers. Normal lumbar range of motion include 60 degrees of flexion, 25 degrees of extension, and 25 degrees of lateral bending
Level of Functional Disability | Functional Disability will be recorded as baseline at the time of recruitment and change in score of functional disability will be recorded at the end of 3rd week of treatment.
  Functional Disability will be measured with the Modified Low Back Pain Disability Questionnaire. The scores range from 0-100% with lower scores meaning less disability.
Change in Fear Avoidance Beliefs | Fear Avoidance Beliefs will be observed as baseline at the time of recruitment and any change in Fear Avoidance Beliefs will be observed at the end of 3rd week of treatment.
  Fear Avoidance Beliefs will be observed using Fear Avoidance Beliefs Questionnaire. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Change in Muscle Activation of Lumbar Multifidus (LM) and Transversus Abdominis (TrA) | The Thickness of muscles will be recorded as baseline at the time of recruitment and change in thickness representing activation will be measured at follow up at the end of 3rd week of treatment.
  Muscle Activation of Lumbar Multifidus (LM) and Transversus Abdominis (TrA) will be measured with Rehabilitative Ultrasound Imaging (RUSI).The activation of muscle is represented through change in thickness level of muscle observed through RUSI. The normal thickness of TrA is 3.93mm and LM is 28.99mm.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr Ashfaq Ahmed, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Participants data that underlies the results after de-identification
Supporting Information: Study Protocol
Time Frame: Immediately after publication
Access Criteria: Researchers who provide methodological sound proposal